CLINICAL TRIAL: NCT00743860
Title: A Study to Evaluate the Pharmacokinetics of the Enteric-Coated Micronized Free Base Formulation of Darapladib [SB-480848] and Its Metabolites in Healthy Volunteers.
Brief Title: A Healthy Volunteer Pharmacokinetic Study of Single and Repeat Doses of SB-480848
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPL112498
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerosis
Keywords: darapladib; pharmacokinetics; metabolite; SB-480848
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose (Experimental): single oral dose
  Interventions: Drug: darapladib
- Repeat Dose (Experimental): 28 day repeat dose
  Interventions: Drug: darapladib

INTERVENTIONS:
Drug: darapladib — experimental drug

SUMMARY:
This study is designed to assess the pharmacokinetics of darapladib and its metabolites following single and 28 days of repeat dosing of darapladib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea
* Child-bearing potential and agrees to use one of the contraception methods per protocol for an appropriate period of time prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight >50 kg and BMI within the range 19 - 30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A positive pre-study drug/alcohol screen.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication
* Consumption of grapefruit or grapefruit juice within 7 days prior to first dose of study medication.
* History of drug abuse.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of anaphylaxis, anaphylactoid (resembling anaphylaxis) reactions or severe allergic responses.
* History of cholecystectomy or biliary tract disease, or a history of liver disease with elevated liver function tests of known or unknown etiology.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if heparin is to be used for flushing a cannula).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Use of oral, injected and implanted hormonal methods of contraception for female subjects.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary PK endpoints will include AUC and Cmax of darapladib and its metabolites (M10, M3 and M4) following single and repeat oral doses. Metabolite to parent AUC and Cmax ratio for each metabolite will be calculated as data permit. | following single and 28 day repeat dose
Clinical safety data (spontaneous AE reporting, vital signs, nursing/physician observation, and clinical laboratory tests) will be the primary safety endpoint. | throughout study

SECONDARY OUTCOMES:
Secondary PK endpoints will include Tmax and T½ of darapladib and its metabolites (M10, M3 and M4) as data permit. | following single and 28 day repeat dose
Plasma Lp-PLA2 activity, expressed in terms of percent inhibition relative to baseline, as data permit. | following single and repeat dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: LPL112498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LPL112498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LPL112498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LPL112498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LPL112498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LPL112498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LPL112498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register